CLINICAL TRIAL: NCT04926558
Title: TROMS (Trainee Reported Outcome Measurement): the New Era of Surgical Evaluation
Acronym: TROMS
Status: Recruiting | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Patricia Sanchez Velazquez, Clinical investigator, Hospital del Mar
Other Study IDs: HMar2021
Record Dates: First submitted 2021-03-24; First posted 2021-06-15 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Surgical Procedure, Unspecified
Keywords: TROMS; PROMS; surgical assessment; learning curve; OSATS; MIR

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
TROMS (trainee reported outcome assessment): assessment of surgical training of residents in general surgery

ELIGIBILITY:
Inclusion criteria:

All surgical residents in the department of general and digestive surgery

Exclusion criteria:

Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all surgical residents of HMar
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of surgical skills achieved by residents | 5 years
  Surgical performance will be evaluated in a random assigned operation by mentors using an specific OPRS (Operative Performance Rating System)

SECONDARY OUTCOMES:
Trainee reported outcomes measurements | 5 years
  Using a specific scale, we aim to measure the satisfaction perceived by our surgical residents concerning their training

CONTACTS AND LOCATIONS:
Locations (1):
- Parc de Salut Mar de Barcelona- Hospital del Mar, Barcelona, Catalonia, Spain